CLINICAL TRIAL: NCT01373008
Title: Inhaled Extra-fine Hydrofluoalkane-beclomethasone (QVAR) in Premature Infants With Bronchopulmonary Dysplasia (BPD); Prospective, Double Blind, Randomized Placebo-control, Multi-center Study
Brief Title: Inhaled Extra-fine Hydrofluoalkane-beclomethasone (QVAR) in Premature Infants With Bronchopulmonary Dysplasia (BPD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Schneider Children's Medical Center, Israel (Other); Meir Hospital, Kfar Saba, Israel (Other); Kaplan Medical Center (Other); Barzilai Medical Center (Other); Laniado Hospital (Other); HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0110-10
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Inhaled steroids; bronchopulmonary dysplasia; Infants with moderate to severe BPD
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled QVAR (Experimental): Inhaled QVAR 100 mic via aerochamber twice daily until 3 month post discharge
  Interventions: Drug: Inhaled extra-fine hydrofluoalkane-beclomethasone (QVAR)
- Inhaled placebo (Placebo Comparator): Inhaled nonmedicated MDI [metered dose inhaler] in a similarly marked aerosol chamber using the same delivery technique, obtained from the drug manufacturer
  Interventions: Drug: Inhaled extra-fine hydrofluoalkane-beclomethasone (QVAR)

INTERVENTIONS:
Drug: Inhaled extra-fine hydrofluoalkane-beclomethasone (QVAR) — Infants will be randomized for Inhaled QVAR 100 microgram or placebo twice daily with spontaneous tidal breathing for 30 seconds via aerochamber with face mask for the study period.

SUMMARY:
Premature infants with chronic lung disease (bronchopulmonary dysplasia [BPD]) are commonly treated with inhaled steroids, an optional treatment according to textbooks and guidelines . However, the evidence supporting this treatment in spontaneously breathing infants is limited, and based on only two randomized, placebo-controlled trials (RCT) with relative small number of infants . The Cochrane review concluded that these studies do not allow firm conclusions with regard to the efficacy of inhaled steroids in non-ventilated infants . Thus, there is no doubt that there is a need for more RCT in order to ascertain the role of inhaled steroids in infants with BPD. Because of its physical properties that theoretically make QVAR an attractive therapy in infants and studies showing it to be as effective as and with similar safety profile as other inhaled steroids in children, the investigators hypothesized that inhaled QVAR will be an effective therapy in infants with BPD.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with moderate to severe BPD, defined as oxygen <30%, or >30% or with positive pressure support at 36 weeks corrected gestational age, respectively
2. Parents signed an informed consent
3. The parents will comply with the 3 months study follow-up requirements, as judged by the site principal investigator.

Exclusion Criteria:

1. Congenital malformation
2. Cardiac disease (including active PDA)
3. Intraventricular hemorrhage grade III-IV
4. Unstable conditions such as sepsis, apneas, ets. at time of enrollment.

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be to compare the rate of readmissions to the hospital for BPD exacerbation during the study period between infants treated with QVAR vs. placebo. | 4 months

SECONDARY OUTCOMES:
Clinical outcomes at each visit | 4 months
  During each visit the following parameters will be charted: Date, vital signs (heart rate, respiratory rate, blood pressure, oxygen pulse oximetry) and physical examination (respiratory distress [0-none, 2- mild, 5-severe], wheezing [0-none, 2- mild, 5-severe], crepitations [0-none, 2- mild, 5-severe]). Will check growth, oxygen need, and in some infant adrenal suppression by urine examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel